CLINICAL TRIAL: NCT05378893
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single-and-Multiple-Ascending Subcutaneous Doses of DR10624
Brief Title: A First in Human (FIH) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DR10624
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Doer Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR10624-101
Record Dates: First submitted 2022-03-25; First posted 2022-05-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Healthy, Obesity, Metabolically
MeSH Terms: conditions — Obesity, Metabolically Benign | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single-ascending dose：Part1：DR10624 (Experimental): Escalating doses of DR10624 for injection administered subcutaneously in healthy participants or obese but otherwise healthy participants
  Interventions: Drug: DR10624 for injection
- Single-ascending dose：Part1：placebo (Placebo Comparator): Escalating doses of placebo for injection administered subcutaneously in in healthy participants or obese but otherwise healthy participants
  Interventions: Drug: Placebo
- Multiple-ascending dose：Part2：DR10624 (Experimental): Escalating doses of DR10624 for injection administered subcutaneously in obese adult subjects with moderate hypertriglyceridemia
  Interventions: Drug: DR10624 for injection
- Multiple-ascending dose：Part2：placebo (Placebo Comparator): Escalating doses of placebo for injection administered subcutaneously in obese adult subjects with moderate hypertriglyceridemia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DR10624 for injection — administered via subcutaneous injection
  Arms: Multiple-ascending dose：Part2：DR10624; Single-ascending dose：Part1：DR10624
Drug: Placebo — administered via subcutaneous injection
  Arms: Multiple-ascending dose：Part2：placebo; Single-ascending dose：Part1：placebo

SUMMARY:
DR10624 is an Fc fusion protein tri-agonist with balanced glucagon-like peptide-1 receptor (GLP-1R)/glucagon receptor (GCGR)/ fibroblast growth factor 21 receptor (FGF21R) agonizing activities. The objectives of the planned clinical investigation will be to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single- and multiple-ascending doses of DR10624 via subcutaneous (SubQ) injection in a randomized, placebo-controlled, double-blind study.

DETAILED DESCRIPTION:
This study includes 2 parts( 1 and 2). Part 1 involves a single dose of DR10624 taken as a subcutaneous injection just under the skin. Part 2 involve multiple doses of DR10624 taken as a subcutaneous injection (SC) just under the skin. Each participant will enroll in only one part.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.
2. Female subjects (heterosexually active, of childbearing potential, not pregnant, not trying to become pregnant, and not lactating) are eligible to participate if they agree to total abstinence from heterosexual intercourse or use a highly effective method of birth control listed below, from screening through until at least 30 days after the last dose of the study drug.

   Male subjects with female partners of childbearing potential are eligible to participate if they are vasectomized, or agree to total abstinence from heterosexual intercourse, from screening through until at least 30 days after the last study dose, or use of an effective method of birth control listed above, from screening through until at least 30 days after the last study dose. Male subjects must refrain from sperm donation throughout the study and for 30 days after the last study dose.
3. The subject agrees to comply with all protocol requirements.
4. The subject is able to provide written informed consent.

Additional inclusion criteria for Part 1:

1. The subject is male or female 18 to 55 years of age, inclusive.
2. The subject has a body weight ≥50 kg at screening and a BMI of 18 to 32 kg/m2, inclusive, or.
3. The subject has a BMI of 30 to 40 kg/m2, inclusive, at screening in obesity subjects cohort.

Additional inclusion criteria for Part 2:

1. The subject is male or female 18 to 60 years of age, inclusive.
2. The subject has a BMI of 30 to 45 kg/m2 at screening, inclusive.
3. Fasting triglyceride ≥150 mg/dL (1.7 mmol/L), and <500 mg/dL (5.7 mmol/L), at screening.

Exclusion Criteria:

1. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
2. The subject has a personal or family history of medullary thyroid cancer, or multiple endocrine neoplasia syndrome Type 2, or a screening calcitonin ≥50 ng/L.
3. The subject has a history of chronic pancreatitis or episode of acute pancreatitis within 3 months of screening.
4. In Part 1, the subject has used any prescription medications (excluding oral contraceptives, paracetamol, and ibuprofen) within 14 days before the first dose of study drug. In Part 2, the subjects have been on stable lipid-lowering therapy <8 weeks before the first dose of study drug.
5. The subject has consumed alcohol within 48 hours before dosing or during the confinement period.
6. The subject is a smoker or has used tobacco, nicotine, or nicotine-containing products.
7. The subject has a history of alcohol abuse or drug addiction within the last year or excessive alcohol consumption.
8. The subject has a positive test result for drugs of abuse and/or alcohol abuse at screening and check-in for the first inpatient period.
9. The subject is involved in strenuous activity or contact sports within 48 hours before admission.
10. The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
11. The subject has total cholesterol >10.3 mmol/L or triglycerides ≥5.7 mmol/L (500 mg/dL) at screening.
12. The subject has clinically significant history or presence of ECG findings as determined by the investigator at screening and check-in,

    - Uncontrolled hypertension (defined as systolic blood pressure (SBP) ≥160 mmHg, and/or diastolic blood pressure (DBP) ≥100 mmHg), angina, bradycardia (if assessed as clinically significant by the investigator), or severe peripheral arterial circulatory disorders.
13. The subject has a history of relevant drug and/or food allergies (ie, allergy to DR10624 or excipients, or any significant food allergy that could preclude a standard diet in the clinical unit).
14. The subject has a history of severe allergic or anaphylactic reactions.
15. The subject has experienced a >5% loss in body weight within 2 months prior to screening.
16. Female subjects who are pregnant or lactating.
17. The subject has a positive test for severe acute respiratory syndrome corona virus 2 (SARS-CoV-2). A positive rapid antigen test (RAT), isothermal nucleic acid amplification, or polymerase chain reaction (PCR) coronavirus disease-2019 (COVID-19) test during screening or at admission is acceptable provided the subject has a known previous COVID-19 infection ≥3 weeks prior to dosing, has recovered, and is now asymptomatic
18. The subject has received study drug in another investigational study within 30 days of dosing.
19. In the opinion of the investigator, the subject is not suitable for entry into the study.

Additional exclusion criteria for subjects in Part 2:

1. Subjects with coagulopathies.
2. Poorly controlled diabetes, defined as HbA1c >8.5% at screening.
3. The subject has been treated with the following anti-diabetic agents, glucagon-like peptide-1 receptor agonist (GLP-1Ra), dipeptidyl peptidase-4 inhibitors (DPP-4i), or insulin, within 30 days prior to screening until the follow-up visit.
4. The subjects have >2 × upper limit of normal (ULN) of either alanine aminotransferase (ALT) or aspartate aminotransferase (AST), or >1.5 × ULN for bilirubin or alkaline phosphatase at screening.
5. Subjects with contraindications to MRI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more treatment-emergent adverse event (TEAE), serious adverse event (SAE) and adverse event of special interest (AESI). | baseline through day 29(part 1)or day 106(part 2)
  Number of participants with one or more TEAE, SAE and AESI.

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve (AUC) | baseline through day 29(part 1)or day 106(part 2)
  Area under the serum concentration versus time curve (AUC)
Maximum observed serum concentration (Cmax) | baseline through day 29(part 1)or day 106(part 2)
  Maximum observed serum concentration (Cmax)
Time to reach maximum observed serum concentration (Tmax) | baseline through day 29(part 1)or day 106(part 2)
  Time to reach maximum observed serum concentration (Tmax)
Terminal elimination half-life (t1/2) | baseline through day 29(part 1)or day 106(part 2)
  Terminal elimination half-life (t1/2)
Mean residence time (MRT) | baseline through day 29(part 1)or day 106(part 2)
  Mean residence time (MRT)
Apparent clearance after extravascular administration (CL/F) | baseline through day 29(part 1)or day 106(part 2)
  Apparent clearance after extravascular administration (CL/F)
Apparent volume of distribution during the terminal elimination phase after extravascular administration (Vz/F) | baseline through day 29(part 1)or day 106(part 2)
  Apparent volume of distribution during the terminal elimination phase after extravascular administration (Vz/F)
AUC from time 0 to the time of the dosing interval (AUC0-t) | baseline through day 106(part 2)
  AUC from time 0 to the time of the dosing interval (AUC0-t)
Accumulation ratio (AR) | baseline through day 106(part 2)
  Accumulation ratio (AR)
Predose concentrations(Ctrough) | baseline through day 106(part 2)
  Predose concentrations(Ctrough)
change in body weight | baseline through Day 85
  change in body weight
change in adiponectin | baseline through Day 85
  change in adiponectin
change in BMI | baseline through Day 85
  change in BMI
change in waist circumference | baseline through Day 85
  change in waist circumference
change in fasting lipid profile | baseline through Day 85
  change in fasting lipid profile
change in fasting plasma glucose (FPG) | baseline through Day 85
  change in FPG
change in HbA1c | baseline through Day 85
  change in HbA1c
change in C-peptide | baseline through Day 85
  change in C-peptide
change in fasting insulin | baseline through Day 85
  change in fasting insulin
change in glucagon | baseline through Day 85
  change in glucagon
change in homeostatic model assessment index of insulin resistance (HOMA-IR) and homeostatic model assessment index of beta-cell function (HOMA-B) | baseline through Day 85
  change in HOMA-IR and HOMA-B
change in Partial area glucose level versus time curve from time 0 to 4 hours (△AUC0-4h) | baseline through Day 85
  change in Partial area glucose levels versus time curve from time 0 to 4 hours (△AUC0-4h)
change in Partial area insulin level versus time curve from time 0 to 4 hours (△AUC0-4h) | baseline through Day 85
  change in Partial area insulin levels versus time curve from time 0 to 4 hours (△AUC0-4h)
change in Partial area C-peptide level versus time curve from time 0 to 4 hours (△AUC0-4h) | baseline through Day 85
  change in Partial area C-peptide levels versus time curve from time 0 to 4 hours (△AUC0-4h)
change in Partial area glucagon level versus time curve from time 0 to 4 hours (△AUC0-4h) | baseline through Day 85
  change in Partial area glucagon levels versus time curve from time 0 to 4 hours (△AUC0-4h)
change percentage of time spent of glucose in target range 3.9 to 10 mmol/L (TIR), time above target range (TAR), time below target range (TBR), 24-hour mean glucose, and glucose variability | baseline through Day 85
  change in TIR, TAR, TBR, 24-hour mean glucose, and glucose variability
change in hepatic fat fraction measured by magnetic resonance imaging-proton density fat fraction (MRI-PDFF ) in part 2 | baseline through Day 85
  change in hepatic fat fraction measured by MRI-PDFF in part 2
Change in liver stiffness by FibroScan in subjects with baseline hepatic fat of at least 8% | baseline through Day 85
  Change in liver stiffness by FibroScan in subjects with baseline hepatic fat of at least 8%
Change in the liver function parameters (ALT, AST, alkaline phosphatase (ALP), and gamma-glutamyltransferase (GGT)) | baseline through Day 85
  Change in the liver function (ALT, AST, alkaline phosphatase (ALP), and gamma-glutamyltransferase (GGT))
Change in Fibrosis 4 score (FIB-4) and non-alcoholic fatty liver disease fibrosis score (NFS) | baseline through Day 85
  Change in FIB-4 and NFS

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Cole, DHPharm, Principal Investigator — New Zealand Clinical Research (NZCR); Yanshan Huang, PhD, Study Chair — Zhejiang Doer Biologics Co., Ltd.; Yongliang Fang, PhD, Study Director — Zhejiang Doer Biologics Co., Ltd.; Junfang Xu, MD, Study Director — Huadong Medicine Co., Ltd.
Locations (1):
- New Zealand Clinical Research, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: No